CLINICAL TRIAL: NCT07270549
Title: GAIN-CTNNB1: A Phase I/II Open-Label Trial To Evaluate the Safety, Tolerability, and Preliminary Efficacy of Intracerebroventricular Administration of an AAV9 Based Gene Replacement Therapy in Paediatric Patients With CTNNB1 Neurodevelopmental Syndrome
Brief Title: Gene Replacement Therapy for Treatment of Paediatric Patients With CTNNB1 Neurodevelopmental Syndrome
Acronym: GAIN-CTNNB1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CTNNB1 Foundation (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Damjan Osredkar, Prof. Damjan Osredkar, MD, PhD, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0120-536/2025-2711; 2025-522719-40-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: CTNNB1 Neurodevelopmental Syndrome
Keywords: CTNNB1 neurodevelopmental syndrome; AAV9 mediated gene replacement therapy; Gene replacement therapy; Gene addition therapy; Gene therapy; Clinical trial
MeSH Terms: interventions — Sirolimus; Methylprednisolone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Urbagen, an AAV-9 mediated gene addition therapy
  Interventions: Biological: Urbagen gene addition therapy; Drug: Sirolimus; Drug: Methylprednisolone (Corticosteroid)

INTERVENTIONS:
Biological: Urbagen gene addition therapy — Urbagen is a non-replicating single-stranded adeno-associated viral vector 9 encoding for the human β-catenin protein (AAV9/hCTNNB1 vector). It is administered as a single bilateral ICV infusion.
Drug: Sirolimus — The use of sirolimus will be consistent with other AAV-9 gene therapy protocols. On Day -7 prior to the administration of URBAGEN, participants will receive a loading dose of sirolimus (3 doses of 1 mg/m2 every four hours). The following day, participants will begin a maintenance dose of sirolimus (0,5 mg/m2/day in 2 divided doses daily), which they will continue for a minimum of 10 months.
Drug: Methylprednisolone (Corticosteroid) — The use of methylprednisolone will be consistent with other AAV-9 gene therapy protocols. On the day of dosing (Day 0), participants will receive a dose of IV methylprednisolone (10 mg/kg to a maximum single dose of 500 mg, infused over 30 minutes). On Day -1 prior to administration of URBAGEN, participants will begin a course of oral prednisolone (1,0 mg/kg/day, maximum dose 30 mg daily). Prednisolone administration will continue for a minimum of four months, followed by a gradual tapering schedule.

SUMMARY:
The goal of this first in human, phase I/II clinical trial is to evaulate the safety, tolerability, and preliminary efficacy of AAV9 mediated gene replacement therapy (Urbagen) in paediatric patients with CTNNB1 neurodevelopmental disorder. The main questions it aims to answer are:

* Is the gene therapy with Urbagen safe and well tolerated?
* Does the gene therapy improve motor function, cognitive function, behavior, sleep, and/or quality of life?

Participants will:

* Undergo screening assessments to ensure eligibility.
* Recieve a single dose of gene therapy via bilateral intracerebroventricular administration.
* Recieve prophylactic immunosuppresants (methylprednisolone, sirolimus).
* Attend follow-up visits for safety monitoring and clinical assessments over the course of three years.

DETAILED DESCRIPTION:
CTNNB1 syndrome is a severe monogenic neurodevelopmental disorder caused by de novo mutations in the CTNNB1 gene. It presents with global developmental delay, spastic dystonic motor impairment, intellectual disability, absent or minimal speech, and a high prevalence of autistic traits.

Urbagen is an investigational gene addition therapy designed to restore functional CTNNB1 expression and improve neurological and developmental outcomes in affected patients. It is a recombinant, single-stranded adeno-associated viral vector serotype 9 (AAV9) encoding the human CTNNB1 gene under the control of the cytomegalovirus enhancer/chicken-β actin hybrid (CBh) promoter. The AAV9 vector facilitates targeted delivery to the central nervous system (CNS), crossing the blood-brain barrier (BBB) and ensuring localized gene expression to address the neurological deficits associated with CTNNB1 syndrome. The therapy is designed as a single-dose bilateral intracerebroventricular (ICV) infusion. The ICV route was selected based on its ability to achieve widespread CNS transduction while minimizing peripheral exposure, as demonstrated in preclinical models.

The goal of this first in human, phase I/II clinical trial to establish the safety, tolerability, and preliminary efficacy of AAV9 mediated gene replacement therapy (Urbagen) in paediatric patients with CTNNB1 syndrome. Urbagen has received orphan drug designation by European Medicines Agency (EMA). The clinical trial was approved by EMA/JAZMP.

This is a monocentric trial conducted at the University Children's Hospital, University Medical Centre Ljubljana, Slovenia. Twelve international participants will receive a single dose of Urbagen via bilateral intracerebroventricular administration. Prophylactic immunosuppresants (methylprednisolone, sirolimus) will be used to reduce the risks of immune-mediated complicationts. Participants will be assessed with a variety of tests during the screening and follow-up period with a total follow up of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant aged 2-12 years at the time of informed consent (Part A: 6-12 years, Part B: 2-12 years).
* Child aged 4 to 12 years has to weigh at least 13,3 kg: 5,0E+14 vg.
* Child aged 3 years has to weigh at least 11,96 kg: 4,5E+14 vg.
* Child aged 2 years has to weigh at least 10,94 kg: 4,11E+14 vg.
* Genetically confirmed diagnosis of CTNNB1 syndrome with a heterozygous pathogenic or likely pathogenic variant in the CTNNB1 gene (Class 4/5 according to American College of Medical Genetics and Genomics), confirmed by geneticist at screening.
* Informed consent from the parents/legal guardians of the participant.
* Parents/legal guardians are willing and able to comply with all protocol visits and procedures.
* Parents/legal guardians are willing and able to reside within 1 hour of the site at which the clinical trial will be conducted for at least 4 months post-dosing. Parents/legal guardians will be informed that this period may be increased in the case of a safety event or concern.
* Parents/legal guardians must agree for the participant not to participate in any other interventional study whilst enrolled in this clinical trial.
* Investigator will check vaccination status of each participant and evaluate and confirm its appropriateness per age and participant's home country. The last vaccination dose must be received a minimum of 30 days prior to the start of immunosuppressants.
* Female participants who are post-menarcheal must have a negative urine pregnancy test at screening and and be willing to have additional pregnancy tests during the study.
* Participant's parents/legal guardians must agree to refrain from future donation of the participant's blood, blood products, tissue, and organs after receiving the IMP due to theoretical risks associated with AAV genome persistence in tissues.
* Participant's use of concomitant medications must be stable for at least 28 days prior to IMP dosing.

Exclusion Criteria:

* Participant has a mutation in the CTNNB1 gene which is predicted to result in a gain-of-function effect (e.g. p.G575R) or dominant negative effect (e.g. p.Y333*, p.Q193*, p.A317Vfs8* and p.S352fs*) on the Wnt/β-catenin pathway, or any variant that, in the opinion of the PI, is inconsistent with the mechanism of action of the gene replacement therapy.
* Participant has a concomitant genetic diagnosis or neurodevelopmental syndrome that in the opinion of the investigator could interfere with safety, ability to perform assessments, or data interpretation.
* Participant tests positive for AAV9 antibody with titers >1:50 for AAV9 antibodies utilizing an enzyme linked immunospot.
* Participant has a known allergy or hypersensitivity to any ingredients or excipients of the IMP, or to immunosuppressants or pre-medications specified within the trial protocol.
* Participant with a history of receiving immune-modulating agents (such as chemotherapy, radiotherapy, intravenous steroids, other immunosuppressive agents) within 3 months prior to dosing. Topical or inhaled corticosteroid treatment may be permitted at the discretion of the investigator.
* Participant has a significant concurrent illness or infection within 30 days prior to dosing which could compromise safety.
* Participant screens positive for acute Coronavirus disease 2019 (COVID-19), confirmed with PCR from a pharyngeal swab sample.
* Participant has serologic evidence of current human immunodeficiency virus (HIV)-1 or HIV-2 infection.
* Participant has acute or chronic hepatitis B or C infections, including:

  * Serologic evidence of hepatitis C infection (positive core antibody)
  * Serologic evidence of acute or chronic active hepatitis B (positive core antibody and/or positive surface antigen)
* Participant diagnosed with a concomitant neurodevelopmental disorder unrelated to CTNNB1.
* Participant with congenital malformation(s) significantly affecting the nervous system.
* Participant with a history of traumatic, metabolic, vascular or infective brain injury with persistent neurological deficits per investigator's judgement.
* Participant has contraindications for MRI brain.
* Participant has a clinically significant increase in seizure frequency as determined by the investigator or clinically documented episode of generalized status epilepticus (≥30 minute generalized tonic-clonic seizure) within 4 weeks of the baseline visit.
* Participant has severe contractures, as determined by the investigator at screening, which are considered likely to interfere with their ability to complete assessments of motor function.
* Participant has increased intracranial pressure, tumor, vascular abnormality, or any major structural anomaly which could complicate or increase the risk of ICV administration of the IMP. Or the participant has any other contraindication to the ICV procedure.
* Participant has a significant congenital cardiac defect that according to the investigator represents a significant safety risk.
* Participant has a left ventricular ejection fraction (LVEF) < 50% on echocardiogram on previous assessment or at screening.
* Participants with clinically significant cardiovascular abnormalities, including clinically significantly prolonged QT interval in ECG (QT interval corrected using Fridericia's formula (QTcF) ≥ 450 ms at screening).
* Participant is assessed as being unable to tolerate anesthesia required for ICV administration and/or sedation required for other study procedures.
* Participant requiring invasive ventilatory support (e.g. endotracheal ventilation or tracheostomy) within the 6 months prior to enrolment.
* Participant has clinically significant liver disease, defined as any of:

  * Aspartate aminotransferase >3,0 x ULN (Grade 1 CTCAE v5.0)
  * Alanine aminotransferase >3,0 x ULN (Grade 1 CTCAE v5.0)
  * Gamma-glutamyl transferase >2,5 x ULN (Grade 1 CTCAE v5.0)
  * Bilirubin >1,5 x ULN (Grade 1 CTCAE v5.0)
* Clinically significant structural abnormality on liver ultrasound.
* Participant has clinically significant renal disease or impairment that could affect safety:

  * Creatinine (>1,5 ULN) (Grade 1 CTCAE v5.0)
  * GFR <50% LLN (Grade 1 CTCAE v5.0)
* Clinically significant structural abnormality on kidney ultrasound.
* Participant has any of the following abnormal, clinically significant laboratory test results during screening. A single repeat will be permitted.

  * Significant thrombocytopenia (Platelet count <150 x 109/L)
  * Neutropenia (Absolute neutrophil count <1 x 109/L)
  * Persistent leukopenia: <2 x 109/L or leukocytosis: >20 x 109/L
  * Significant anemia (hemoglobin <100 g/L)
  * Abnormal coagulation (prothrombin time or partial thromboplastin time above ULN)
* Participant has a history of a biopsy-confirmed malignancy.
* Participant has a history of major surgery within six months prior to enrolment or planned surgery during first 12 months of study.
* Participant has any other significant concomitant medical disorder which could confound the interpretation of safety or efficacy data as determined by PI or medical monitor.
* Participant has been enrolled in another interventional clinical trial within 1 year prior to enrolment.
* Participant has previously received gene or cell therapy.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Assesing safety and tolerability of Urbagen. | 5 years (multiple timepoints)
  Monitoring for any adverse events and serious adverse events in all participants.

SECONDARY OUTCOMES:
Improvement in motor function as measured by the Bayley Scale of Infant Development 4. | 5 years (multiple timepoints)
Improvement in motor function as measured by the Wearable Syde Device (in ambulant patients). | 5 years (multiple timepoints)
Improvement in dystonia as measured by the Burke-Fahn-Marsden Dystonia Rating Scale. | 5 years (multiple timepoints)
Improvement in spasticity as measured by the 13-item Spastic Paraplegia Rating Scale. | 5 years (multiple timepoints)
Improvement in cognitive function as measured by the Bayley Scale of Infant Development 4. | 5 years (multiple timepoints)
Improvement in cognitive function as measured by the Vineland Adaptive Infant Behavior Scale 3. | 5 years (multiple timepoints)
Improvement in cognitive function as measured by the Wechsler Non-Verbal Intelligence Scale. | 5 years (multiple timepoints)
Improvement in communication as measured by the Vineland Adaptive Scale 3. | 5 years (multiple timepoints)
Behavioral Improvement measured by the Aberrant Behavior Checklist. | 5 years (multiple timepoints)
Behavioral Improvement measured by the M-CHAT or Autism Spectrum Quotient (depending on the participant's age). | 5 years (multiple timepoints)
Improvement in sleep as measured by the Bruni Sleep Disturbance Scale. | 5 years (multiple timepoints)
Improvement in epilepsy as measured by seizure frequency. | 5 years (multiple timepoints)
Improvement in Quality of Life as measured by Pediatric QOL Inventory - Family and Core module (age appropriate). | 5 years (multiple timepoints)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zakelj N, Gosar D, Mirosevic S, Sanders SJ, Ljungdahl A, Kohani S, Huang S, Leong LI, An Y, Teo MJ, Moultrie F, Jerala R, Lainscek D, Forstneric V, Susjan P, Lisowski L, Perez-Iturralde A, Mrak JO, Chan HYE, Osredkar D. Genotypic, functional, and phenotypic characterization in CTNNB1 neurodevelopmental syndrome. HGG Adv. 2025 Oct 9;6(4):100483. doi: 10.1016/j.xhgg.2025.100483. Epub 2025 Jul 18. PMID 40684264
- [Background] Mirosevic S, Khandelwal S, Amerson E, Parks E, Parks M, Cochran L, Gonzalez Hernandez A, Ferraro M, Lisowski L, Perez-Iturralde A, Chung W, Jacob MH, Zakelj N, Lainscek D, Forstneric V, Susjan P, Maruna M, Jerala R, Osredkar D. Paving the way toward treatment solutions for CTNNB1 syndrome: a patient organization perspective. Ther Adv Rare Dis. 2025 Feb 12;6:26330040251318355. doi: 10.1177/26330040251318355. eCollection 2025 Jan-Dec. PMID 39949392
- [Background] Mirosevic S, Khandelwal S, Susjan P, Zakelj N, Gosar D, Forstneric V, Lainscek D, Jerala R, Osredkar D. Correlation between Phenotype and Genotype in CTNNB1 Syndrome: A Systematic Review of the Literature. Int J Mol Sci. 2022 Oct 19;23(20):12564. doi: 10.3390/ijms232012564. PMID 36293418
- [Background] Parichha A, Datta D, Singh A, Talwar I, Yadav S, Bose M, Suresh V, Mirosevic S, Zakelj N, Gosar D, Osredkar D, Tole S. An evolutionarily conserved role for CTNNB1/beta-CATENIN in regulating the development of the corpus callosum. iScience. 2025 Aug 9;28(9):113335. doi: 10.1016/j.isci.2025.113335. eCollection 2025 Sep 19. PMID 40894864
- [Background] Arkar Silan U, Trebse A, Kovac J, Rogac M, Troha Gergeli A, Sket R, Bregant T, Neubauer D, Peterlin B, Osredkar D. Unravelling genetic etiology of cerebral palsy: findings from a Slovenian pediatric cohort. Front Neurol. 2025 Jul 23;16:1615449. doi: 10.3389/fneur.2025.1615449. eCollection 2025. PMID 40771987
- [Background] Groselj U, Kavcic M, Drole Torkar A, Kafol J, Lainscek D, Jerala R, Sever M, Zver S, Sersa G, Cemazar M, Strojan P, Groselj A, Zerjav Tansek M, Mirosevic S, Ivancan S, Prelog T, Gosar D, Orazem Mrak J, Mlinaric M, Bertok S, Kovac J, Kodric J, Battelino S, Pokorn M, Ihan A, Jazbec J, Battelino T, Osredkar D. Gene therapy of rare diseases as a milestone in medicine - overview of the field and report on initial experiences in Slovenia. Orphanet J Rare Dis. 2025 Jun 5;20(1):279. doi: 10.1186/s13023-025-03828-8. PMID 40474241
- See also: CTNNB1 Foundation — https://ctnnb1-foundation.org/